CLINICAL TRIAL: NCT02745808
Title: Injectable Collagen Scaffold™ Combined With Human Umbilical Cord-derived Mesenchymal Stem Cells (HUC-MSCs) for the Improvement of Erectile Function in Men With Diabetes
Brief Title: Injectable Collagen Scaffold™ Combined With HUC-MSCs for the Improvement of Erectile Function in Men With Diabetes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAS-XDA-DEF/IGDB
Record Dates: First submitted 2016-04-12; First posted 2016-04-20 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2016-04

CONDITIONS: Erectile Dysfunction; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HUC-MSCs (Experimental): Intracavernous injection of 15 million HUC-MSCs.
  Interventions: Biological: HUC-MSCs
- Injectable Collagen Scaffold + HUC-MSCs (Experimental): Intracavernous injection of injectable collagen scaffold combined with 15 million HUC-MSCs.
  Interventions: Biological: Injectable Collagen Scaffold + HUC-MSCs

INTERVENTIONS:
Biological: HUC-MSCs — The subjects will receive intracavernous injection of HUCMSC.
  Arms: HUC-MSCs
Biological: Injectable Collagen Scaffold + HUC-MSCs — The subjects will receive intracavernous injection of the mixture of injectable collagen scaffold and HUC-MSCs.
  Arms: Injectable Collagen Scaffold + HUC-MSCs

SUMMARY:
The intent of this clinical study is to answer the questions: 1) is the proposed treatment feasible; 2) is treatment effective in improving the disease pathology of patients with diagnosed diabetic erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or 2 diabetes,blood glucose controlled well, no effective with oral PDE-5i
2. Have a consistent partner who is willing to engage in sexual activity more than twice per month during the study
3. Males, age 20-65 years
4. IIEF-5 score is under 16
5. Penile arterial insufficiency or venous leakage (doppler): peak systolic velocity（PSV） <25 cm/sec, or peak systolic velocity（PSV）>25 cm/sec, end-diastolic velocity（EDV）> 5cm/sec, resistance index（RI）<0.75
6. HbA1c is between 6.5%-10%
7. Physical examination with no abnormalities
8. Willing to consent to participate in the study follow-up
9. Willing to limit alcohol intake eliminate use of recreational drugs for sexual encounters.

Exclusion Criteria:

1. Severe cardiovascular disease (angina, arrhythmia, cardiac failure, stroke), kidney failure, respiratory failure; history of malignancy
2. Positive for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) syphilis test
3. Testosterone level is less than 200ng/dL
4. Serum AST/ALT >3*upper limit of normal or creatinine >1.5*upper limit of normal
5. HbA1c exhibit greater than 10%
6. In the investigators judgment, with clinical significance of penis abnormalities, or has received penile prosthesis implantation surgery
7. Patients partner is trying to conceive during the trial period
8. Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study
9. Unwilling and/or not able to give written informed consent

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability assessed by Adverse Events | 1 month after intervention

SECONDARY OUTCOMES:
Improvement in IIEF-5 (International Index of Erectile Function) | 1,3,6,9 and 12 months
  The subjects must fill in the questionnaire of IIEF-5 every visit to evaluate erectile function
Improvement in penile colour Doppler ultrasonography | 1,3,6,9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China